CLINICAL TRIAL: NCT00996853
Title: Post-Authorization Safety Study (PASS) of GlaxoSmithKline Biologicals' Pandemic Influenza Vaccine (GSK2340272A) in the United Kingdom (UK)
Brief Title: Post-Authorization Safety Study of GSK Biologicals' Pandemic Influenza Vaccine (H1N1) in the United Kingdom
Acronym: H1N1 PASS UK
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113585
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Influenza
Keywords: safety; Influenza; vaccine; reactogenicity; swine flu
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Total vaccinated cohort: The Total vaccinated cohort will include all subjects with at least one vaccine administration documented.
  Interventions: Other: Safety follow up

INTERVENTIONS:
Other: Safety follow up — Collection of reactogenicity data from diary cards, reporting of medically-attended adverse events, reporting of serious adverse events and adverse events of special interest, reporting of pregnancy outcomes and fatalities.

SUMMARY:
The focus of this study is to assess the safety of GSK's H1N1 vaccine in real life conditions as soon as the vaccine is used, in a mass vaccination programme, and with a system for rapid generation, communication and evaluation of safety data.

This study is a commitment to the European Medicines Agency (EMEA), as part of GlaxoSmithKline Biologicals' (GSK Biologicals') risk management plan for pandemic influenza vaccination.

DETAILED DESCRIPTION:
Collaborator: Medicines and Healthcare products Regulatory Agency

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, and assent where appropriate, obtained from the subject/from the subject's parent(s)/ Legally Acceptable Representative(s) (LAR).
* A male or female subject vaccinated with a first dose of GSK Biologicals' H1N1 pandemic influenza vaccine
* shortly (<24h) before being recruited in the study, and
* within a GP practice participating in the study and where the subject is registered.
* Subjects who the Investigator believes that they and/or their parent(s)/LAR can and will comply with the requirements of the protocol

Exclusion Criteria:

* Subjects already vaccinated with any other H1N1 pandemic vaccine before study enrolment.
* Child in care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population studied will include individuals in priority groups currently considered for H1N1 pandemic vaccination. Subjects not pertaining to these priority groups can also be enrolled.
Sampling Method: Probability Sample
Enrollment: 9206 (Actual)
Dates: Start 2009-10-31 (Actual); Primary Completion 2010-10-20 (Actual); Study Completion 2011-04-06 (Actual)

PRIMARY OUTCOMES:
Medically-attended adverse events | Within one month after any dose

SECONDARY OUTCOMES:
Adverse events solicited to assess reactogenicity | Within seven days after any dose
Serious adverse events and adverse events of special interest | Within six months after the second vaccine dose or within a maximum of eight months after the first dose
Pregnancy outcomes | Within two months after vaccination (last menstrual period up to 45 days after any dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (87):
- United Kingdom (87):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Watford, Hertfordshire
  - GSK Investigational Site, Canterbury, Kent
  - GSK Investigational Site, Blackburn, Lancashire
  - GSK Investigational Site, Wellingborough, Northamptonshire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Frome, Somerset
  - GSK Investigational Site, Addlestone,Surrey
  - GSK Investigational Site, Attleborough, Norfolk
  - GSK Investigational Site, Axbridge, Somerset
  - GSK Investigational Site, Baldock, Herts
  - GSK Investigational Site, Balham, London
  - GSK Investigational Site, Bath, Avon
  - GSK Investigational Site, Bedwell Crescent, Stevenage
  - GSK Investigational Site, Blenheim Walk, Leeds
  - GSK Investigational Site, Botesdale
  - GSK Investigational Site, Boughton, King's Lynn
  - GSK Investigational Site, Bristol, Avon
  - GSK Investigational Site, Bromsgrove,Worcestershire
  - GSK Investigational Site, Chard, Somerset
  - GSK Investigational Site, Chesterfield
  - GSK Investigational Site, Colchester,Essex
  - GSK Investigational Site, Comberton,Cambridge
  - GSK Investigational Site, Darlington, Co. Durham
  - GSK Investigational Site, Devon
  - GSK Investigational Site, Didcot,Oxfordshire
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Ecclesfield
  - GSK Investigational Site, Ellesmere Port,Cheshire
  - GSK Investigational Site, Escrick, York
  - GSK Investigational Site, Essex
  - GSK Investigational Site, Fleetwood
  - GSK Investigational Site, Gosport
  - GSK Investigational Site, Hanworth, Feltham
  - GSK Investigational Site, Harrogate
  - GSK Investigational Site, Harwood, Bolton
  - GSK Investigational Site, Hertfordshire
  - GSK Investigational Site, High Kelling,Holt,Norfolk
  - GSK Investigational Site, Honiton,Devon
  - GSK Investigational Site, Hoyland, Barnsley
  - GSK Investigational Site, Hurstpierpoint, West Sussex
  - GSK Investigational Site, Kent, Sevenoaks
  - GSK Investigational Site, Kettering,Kettering
  - GSK Investigational Site, Kippax,Leeds
  - GSK Investigational Site, Lambeth, London
  - GSK Investigational Site, Lancashire
  - GSK Investigational Site, Lancaster
  - GSK Investigational Site, Langport, Somerset
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Lichfield
  - GSK Investigational Site, London
  - GSK Investigational Site, Lutterworth, Leicestershire
  - GSK Investigational Site, Mossley, Ashton Under Lyne
  - GSK Investigational Site, Nantwich, Cheshire
  - GSK Investigational Site, Norwich, Norfolk
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Orton Goldhay, Peterborough
  - GSK Investigational Site, Oxfordshire
  - GSK Investigational Site, Paiginton, Devon
  - GSK Investigational Site, Radstock, Bath
  - GSK Investigational Site, Romsey, Hampshire
  - GSK Investigational Site, Rowlands Castle
  - GSK Investigational Site, Ruislip
  - GSK Investigational Site, Runcorn, Cheshire
  - GSK Investigational Site, Salisbury, Hampshire
  - GSK Investigational Site, Sedgefield
  - GSK Investigational Site, Shipston-on-Stour, Warwickshire
  - GSK Investigational Site, Somerset
  - GSK Investigational Site, Southbourne, Hampshire
  - GSK Investigational Site, Southsea, Hampshire
  - GSK Investigational Site, Stowmarket,Suffolk
  - GSK Investigational Site, Sunderland
  - GSK Investigational Site, Sway, Hampshire
  - GSK Investigational Site, Swindon, Wiltshire
  - GSK Investigational Site, Tadworth,Surrey
  - GSK Investigational Site, Tarporley,Cheshire
  - GSK Investigational Site, Thornbury, Bristol
  - GSK Investigational Site, Wandsford, Peterborough
  - GSK Investigational Site, Wantage
  - GSK Investigational Site, Wantage, Oxon
  - GSK Investigational Site, Western Approach,Plymouth
  - GSK Investigational Site, Westhoughton, Bolton
  - GSK Investigational Site, Wiltshire, Westbury
  - GSK Investigational Site, Wiltshire
  - GSK Investigational Site, Windemere,Cumbria
  - GSK Investigational Site, Wokingham, Berkshire
  - GSK Investigational Site, York

REFERENCES:
- [Background] Nazareth I, Tavares F, Rosillon D, Haguinet F, Bauchau V. Safety of AS03-adjuvanted split-virion H1N1 (2009) pandemic influenza vaccine: a prospective cohort study. BMJ Open. 2013 Feb 5;3(2):e001912. doi: 10.1136/bmjopen-2012-001912. Print 2013. PMID 23388195
- [Background] Tavares F, Nazareth I, Monegal JS, Kolte I, Verstraeten T, Bauchau V. Pregnancy and safety outcomes in women vaccinated with an AS03-adjuvanted split virion H1N1 (2009) pandemic influenza vaccine during pregnancy: a prospective cohort study. Vaccine. 2011 Aug 26;29(37):6358-65. doi: 10.1016/j.vaccine.2011.04.114. Epub 2011 May 17. PMID 21596080